CLINICAL TRIAL: NCT03915184
Title: Open Label, Multi-center, Phase 1b/2 Clinical Trial to Evaluate the Safety and Efficacy of Autologous CAR BCMA T Cells (CT053) in Patients With Relapsed and/or Refractory Multiple Myeloma (LUMMICAR STUDY 2)
Brief Title: Clinical Trial to Evaluate Zevor-cel (CT053) in Patients With Relapsed and/or Refractory Multiple Myeloma (LUMMICAR STUDY 2)
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: CARsgen Therapeutics Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CT053-MM-02 (LUMMICAR STUDY 2)
Record Dates: First submitted 2019-04-03; First posted 2019-04-16 (Actual); Last update posted 2023-12-19 (Actual); Status verified 2023-12

CONDITIONS: Multiple Myeloma
Keywords: CAR-T; Carcinoma; Carcinoma, Multiple Myeloma; CT053; zevor-cel
MeSH Terms: conditions — Multiple Myeloma; Carcinoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- CAR-BCMA T Cells (Experimental): Phase 1b will include a dose escalation followed by an expansion cohort to determine the recommended dose for the expansion part. After recommended Phase 2 is determined, patients in Phase 2 will be treated.
  Interventions: Biological: zevor-cel

INTERVENTIONS:
Biological: zevor-cel — A single autologous chimeric antigen receptor-B-cell maturation antigen (CAR-BCMA T cell) infusion
  Other Names: CAR-BCMA T Cell Infusion

SUMMARY:
A phase 1b/2, open label, multi-center, Clinical Study of Chimeric Antigen Receptor T Cells targeting BCMA in patients with relapsed and or refractory multiple myeloma.

DETAILED DESCRIPTION:
This is an open label, multi-center, phase 1b/2 clinical trial to evaluate the safety and efficacy of autologous chimeric antigen receptor-B-cell maturation antigen (CAR-BCMA T cell; zevor-cel/CT053) in patients with relapsed and or refractory multiple myeloma.

Phase 1b of the study will be dose escalation followed by an expansion cohort. After recommended Phase 2 dose is identified in Phase 1b, the enrollment of Phase 2 will start. Following consent, enrolled subjects will undergo a leukapheresis procedure to collect autologous mononuclear cells for manufacture of investigational drug product (zevor-cel). Following manufacture of the drug product, subjects will receive lymphodepletion prior to zevor-cel infusion. All subjects who complete the study, as well as those who withdraw from the study after receiving zevor-cel for reasons other than death or meeting the early termination criteria, will be asked to continue to undergo a 15-year long-term follow-up study.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily signed consent;
2. Age of ≥ 18 and < 80 years;
3. Received sufficient prior lines of myeloma therapy;
4. Received treatment with at least one proteasome inhibitor, one IMiD and CD38 anti body.
5. The patient must be refractory to the last line of therapy.
6. The patients should have measurable disease per IMWG definition.
7. Estimated life expectancy > 12 weeks;
8. ECOG performance score 0-1;
9. Patients should have reasonable CBC counts, renal and hepatic functions;
10. Sufficient venous access for leukapheresis collection, and no other contraindications to leukapheresis;
11. Women of childbearing age must undergo a serum pregnancy test with negative results before screening, and are willing to use effective and reliable method of contraception for at least 12 months after T cell infusion;
12. Men must be willing to use effective and reliable method of contraception for at least 12 months after T cell infusion.

Exclusion Criteria:

1. Pregnant or lactating women;
2. HIV, active hepatitis C virus (HCV), or active hepatitis B virus (HBV) infection;
3. Any uncontrolled active infection;
4. AEs from previous treatment that have not recovered;
5. Patients who have had anti-BCMA therapy;
6. Patients who have graft versus host disease (GvHD);
7. Patients have received stem cell transplantation one year before leukapheresis;
8. Patients have received any anti-cancer treatment before leukapheresis;
9. Patients have received steroids before leukapheresis or lymphodepletion;
10. Patients have plasma cell leukemia, Waldenström macroglobulinemia, POEMS (polyneuropathy, organomegaly, endocrinopathy, monoclonal gammopathy, and skin changes) syndrome or clinically significant symptomatic immunoglobulin light chain (AL) amyloidosis with evidence of end-organ damage;
11. Patients have been administered live attenuated vaccine before leukapheresis or lymphodepletion;
12. Patients allergic to Flu, Cy, tocilizumab, dimethyl sulfoxide (DMSO) or zevor-cel CAR BCMA T cell;
13. Patients have clinical significant cardiac conditions that researchers believe that participating in this clinical trial may endanger the health of the patients;
14. Patients have clinical significant pulmonary conditions;
15. Patients are known to have active autoimmune diseases including but not limited to psoriasis, rheumatoid arthritis and other needs of long-term immunosuppressive therapy;
16. Patients with second malignancies in addition to MM are not eligible;
17. Patients have central nervous system (CNS) metastases or CNS involvement;
18. Patients have significant neurologic disorders;
19. Patients are unable or unwilling to comply with the requirements of clinical trial;
20. Patients have received major surgery prior to leukapheresis or prior to lymphodepletion.

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 105 (Estimated)
Dates: Start 2019-09-25 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2034-12-31 (Estimated)

PRIMARY OUTCOMES:
Incidence of Treatment Related adverse events (AEs) | Day 1 - Month 60
  Incidence of Treatment Related AEs, AEs of special interest and serious adverse events (SAEs)
Identification of Maximum Tolerated Dose (MTD) | Day 1 - Month 60
  Incidence of dose-limiting toxicities (DLTs)
Objective response rate | Day 1 - Month 60
  Objective response rate (ORR) per IMWG by IRC read

SECONDARY OUTCOMES:
Evaluate additional clinical efficacy outcomes with zevor-cel treatment in patients with rrMM | Day 1 - Month 60
  Disease-specific response criteria including, but not limited to: complete response (CR), MRD, very good partial response (VGPR), and partial response (PR) according to the International Myeloma Working Group (IMWG) Uniform Response Criteria for Multiple Myeloma, Time to Response, Time to Progression, Progression Free Survival, best response and Overall Survival
Determine the efficacy of zevor-cel treatment in patients with rrMM, by investigator assessment | Day 1 - Month 60
  ORR, DOR, FPS, OS, MRD, time to response, time to progression, best tumor response
Evaluate zevor-cel PK profile | Day 1 - Month 60
  CAR transgene copy number, peak value, AUC, in vivo persistence
Evaluate ADA profile | Day 1 - Month 60
  Percentage of patients with anti-zevor-cel drug antibodies
Evaluate HRQoL in patients with rrMM from baseline up to study completion | Day 1 - Month 60
  Change from baseline in HRQoL as measured by EORTC QLQ-C30 and QLQ-MY20
Evaluate utilization of hospital resources | Day 1 - Month 60
  Duration of hospitalization and ICU

OTHER OUTCOMES:
BCMA bone marrow expression and soluble BCMA expression in blood | Day 1 - Month 60
  Myeloma cell BCMA expression and serum soluble BCMA
Cytokine profiling | Day 1 - Month 60
  cytokine levels (such as IL-6, INF, et al)
zevor-cel product profiling vs clinical safety and efficacy | Day 1 - Month 60
  zevor-cel product characteristics

CONTACTS AND LOCATIONS:
Overall Officials: Shaji Kumar, MD, Principal Investigator — Mayo
Locations (13):
- United States (12):
  - Mayo Clinic Hospital, Phoenix, Arizona
  - UCSF, San Francisco, California
  - Colorado Blood Cancer Institute, Denver, Colorado
  - Moffitt Cancer Center, Tampa, Florida
  - Dana Farber Cancer Center, Boston, Massachusetts
  - Mayo, Rochester, Minnesota
  - TriStar CMC, Nashville, Tennessee
  - UT Southwestern Medical Center, Dallas, Texas
  - MD Anderson, Houston, Texas
  - Methodist Hosptial, Houston, Texas
  - Huntsman Cancer Center, Salt Lake City, Utah
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Princess Margaret Hospital, Toronto, Ontario, Canada